CLINICAL TRIAL: NCT07128615
Title: A Phase I/II, Double-blinded, Randomized, Placebo-Controlled, Dose Selection Study in Adults to Assess the Safety and Immunogenicity of AZD4117 and AZD5315 Vaccines (PANDA)
Brief Title: A Phase I/II Study on Safety AND Immunogenicity of AZD4117 and AZD5315 Vaccines (PANDA)
Acronym: PANDA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Joint Program Executive Office (JPEO) Chemical, Biological, Radiological, and Nuclear Defense (CBRND) Enabling Biotechnologies (EB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D8500C00001
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Influenza A
Keywords: Avian Influenza A; mRNA Vaccine; Pandemic Influenza; VLP; H5N1; H7N9; AstraZeneca

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking will be secured to the syringe after preparation by unblinded personnel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Arm 1: Dosage Level 1 (DL1) of AZD4117 18 to 64 years of age (Experimental): Participants will receive DL1 AZD4117.
  Interventions: Biological: AZD4117
- Arm 2: Dosage Level 2 (DL2) of AZD4117 18 to 64 years of age (Experimental): Participants will receive DL2 AZD4117.
  Interventions: Biological: AZD4117
- Arm 3: DL1 of AZD4117 >= 65 years of age (Experimental): Participants will receive DL1 AZD4117.
  Interventions: Biological: AZD4117
- Arm 4: DL2 of AZD4117 >= 65 years of age (Experimental): Participants will receive DL2 AZD4117.
  Interventions: Biological: AZD4117
- Arm 5: DL1 of AZD5315 18 to 64 years of age (Experimental): Participants will receive DL1 AZD5315.
  Interventions: Biological: AZD5315
- Arm 6: DL2 of AZD5315 18 to 64 years of age (Experimental): Participants will receive DL2 AZD5315.
  Interventions: Biological: AZD5315
- Arm 7: DL1 of AZD5315 >= 65 years of age (Experimental): Participants will receive DL1 AZD5315.
  Interventions: Biological: AZD5315
- Arm 8: DL2 of AZD5315 >= 65 years of age (Experimental): Participants will receive DL2 AZD5315.
  Interventions: Biological: AZD5315
- Arm 9: placebo 18 to 64 years of age (Placebo Comparator): Participants will receive placebo.
  Interventions: Other: Placebo
- Arm 10: placebo >= 65 years of age (Placebo Comparator): Participants will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AZD4117 — Intramuscular (IM) injection
  Arms: Arm 1: Dosage Level 1 (DL1) of AZD4117 18 to 64 years of age; Arm 2: Dosage Level 2 (DL2) of AZD4117 18 to 64 years of age; Arm 3: DL1 of AZD4117 >= 65 years of age; Arm 4: DL2 of AZD4117 >= 65 years of age
Biological: AZD5315 — IM injection
  Arms: Arm 5: DL1 of AZD5315 18 to 64 years of age; Arm 6: DL2 of AZD5315 18 to 64 years of age; Arm 7: DL1 of AZD5315 >= 65 years of age; Arm 8: DL2 of AZD5315 >= 65 years of age
Other: Placebo — IM injection
  Arms: Arm 10: placebo >= 65 years of age; Arm 9: placebo 18 to 64 years of age

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of two investigational vaccines, AZD4117 and AZD5315 to protect against certain strains of avian Influenza A (H5N1 and H7N9 subtypes).

ELIGIBILITY:
Key Inclusion Criteria:

* Adults, ≥ 18 years of age at the time of signing the informed consent
* Participants who are medically stable such that, according to the judgement of the Investigator, hospitalization within the study period is not anticipated and the participant appears likely to be able to remain on study through the end of protocol-specified follow-up. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to enrollment
* Written informed consent and any locally required authorization (eg, HIPAA in the US) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations

Key Exclusion Criteria:

* History of hypersensitivity to any component of the IMP
* History of hypersensitivity to penicillin and its derivatives
* History of severe adverse reaction and/or severe allergic reaction (eg, anaphylaxis associated with a vaccine
* Known or suspected congenital or acquired immunodeficiency
* Abnormal findings on screening laboratory tests
* Previous history of myocarditis, pericarditis, Guillain-Barré syndrome or any other demyelinating condition
* Known or suspected autoimmune conditions as determined by history and/or physical examination
* Receipt of any other type of seasonal influenza vaccination from 14 days before the first dose until 28 days after the administration of the last dose of IMP
* Receipt of an mRNA vaccine within 28 days before administration of IMP
* Receipt or expected receipt of any other type of licensed or investigational vaccine within 28 days prior to Visit 1 (D1) or Visit 5 (D58)
* Receipt of immunoglobulin or blood products within 6 months prior to administration of study intervention or expected receipt during the study
* Receipt of immune-modifying drugs or immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy within 6 months prior to enrollment (or expected receipt during study), or long-term systemic corticosteroid therapy (prednisolone or equivalent at a dose of ≥ 20 mg daily for more than 2 consecutive weeks) within 6 months prior to enrollment or expected receipt during study. Topical/inhaled steroids or short-term oral steroids are permitted
* Participation in another trial, or receiving interventional Study IMP, in the preceding 90 days or expected receipt of another study intervention (or participation in another trial) during the period of study follow-up
* Acute (time-limited) or febrile (temperature ≥ 38.0 °C [100.4 °F]) illness/infection within 3 days of intended IMP administration
* Individuals who have had a previous confirmed or suspected illness from influenza caused by an H5N1 or H7N9 virus
* Individuals who had household contact with and/or intimate exposure to an individual with laboratory confirmed H5N1 infection, exposure to infected household poultry/ wild birds/cattle or contaminated environments with sick and dead poultry or wild birds or cattle, within 60 days prior to enrollment
* Female participants who are pregnant, lactating, or of childbearing potential and not using a highly effective method of contraception or abstinence from at least 4 weeks prior to IMP administration and until at least 6 months after IMP administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with immediate unsolicited adverse events (AE) | Within 30 minutes after dosing
Percentage of participants with injection site and systemic solicited adverse reactions (AR) | Through 7 days after dosing
Percentage of participants with unsolicited AE | Through 28 days after the last dose
Percentage of participants with serious adverse events (SAE) | Through 12 months after the last dose
Percentage of participants with medically attended adverse events (MAAE) | Through 12 months after the last dose
Percentage of participants with adverse events of special interest (AESI) | Through 12 months after the last dose
Proportion of participants achieving ≥ 1:40 HAI titer post-IMP administration | Day 58
  A binary endpoint, defined as ≥ 1:40 HAI titer post-IMP administration.
Proportion of participants achieving seroconversion post-IMP administration | Day 58
  Seroconversion status, defined as either a pre-IMP administration HAI titer < 1:10 and a post-IMP administration HAI titer ≥ 1:40, or a pre-IMP administration titer ≥ 1:10 and 4-fold increase in post-IMP administration titer.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of HAI antibody | Days 1 to 389
Geometric mean fold-rise (GMFR) of HAI antibody titers from baseline | Days 29 to 389
  The fold rise is calculated as the ratio of the post-dose titer to the pre-dose titer.
Proportion of participants achieving a ≥1:40 HAI titer post-IMP administration | Days 29 to 389
  A binary endpoint, defined as ≥ 1:40 HAI titer post-IMP administration.
Proportion of participants achieving seroconversion post-IMP administration | Days 29 to 389
  Seroconversion status, defined as either a pre-IMP administration HAI titer < 1:10 and a post-IMP administration HAI titer ≥ 1:40, or a pre-IMP administration titer ≥ 1:10 and 4-fold increase in post-IMP administration titer.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Research Site, Long Beach, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Hialeah, Florida
  - Research Site, Stockbridge, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lenexa, Kansas
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Cincinnati, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, North Charleston, South Carolina
  - Research Site, Austin, Texas
  - Research Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/